CLINICAL TRIAL: NCT06391125
Title: LIMIT Trial - Lidocaine With Intramuscular Injection of Benzathine Penicillin G for Treponema Pallidum Treatment
Acronym: LIMIT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Joseph Cherabie, Assistant Professor, Washington University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202401099
Record Dates: First submitted 2024-03-20; First posted 2024-04-30 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Syphilis Infection; Benzathine Penicillin Adverse Reaction
Keywords: Syphilis; Syphilis Treatment; Benzathine Penicillin G; Lidocaine
MeSH Terms: conditions — Syphilis | interventions — Saline Solution; Lidocaine

STUDY DESIGN:
Intervention Model Description: double blinded randomized placebo control trial of addition of the effect on pain of the addition of 0.5ml 1% lidocaine solution to prepackaged benzathine Penicillin G injection, compared to addition of 0.5 ml normal saline solution, in adults being treated for syphilis (Treponema pallidum) infections, within the Infectious Diseases Clinic at Washington University in St. Louis.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both participants and clinicians will be blinded to the contents of the syringe. The nurse filling the syringe will assign the syringes randomly to be injected into L or R gluteal muscle and will label them accordingly, logging the designation in a log book that will remain blinded until the analysis portion of the study. The participant will be blinded as they will receive one site of injection with lidocaine and the other with normal saline, serving as their own intervention and control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lidocaine + Benzathine Penicillin G Arm (Experimental): 0.5ml 1% lidocaine solution added to prefilled 1.2 million units Benzathine Pencillin G syringe which will be injected once into the gluteal muscle of the study participant, the side (left or right) to be randomly assigned with the control assigned to the other gluteal muscle.
  Interventions: Drug: Lidocaine
- Normal Saline + Benzthine Penicillin G Arm (Placebo Comparator): 0.5ml normal saline solution added to prefilled 1.2 million units Benzathine Pencillin G syringe which will be injected once into the gluteal muscle of the study participant, the side (left or right) to be randomly assigned with the study arm assigned to the other gluteal muscle.
  Interventions: Drug: normal Saline

INTERVENTIONS:
Drug: normal Saline — 0.5ml normal saline solution added to prefilled 1.2 million units Benzathine Pencillin G syringe
  Arms: Normal Saline + Benzthine Penicillin G Arm
Drug: Lidocaine — 0.5ml 1% lidocaine solution added to prefilled 1.2 million units Benzathine Pencillin G syringe
  Arms: Lidocaine + Benzathine Penicillin G Arm

SUMMARY:
There is evidence to suggest that lidocaine can help reduce the pain associated with intramuscular injections of benzathine penicillin G (BPG) or Bicillin, used to treat syphilis infections. A study published in the Journal of Family Practice in 2001 compared the pain experienced during bicillin injections with and without the use of lidocaine. The study found that patients who received lidocaine injections before receiving bicillin reported significantly less pain compared to those who received bicillin injections without lidocaine. Per the International Union against Sexually Transmitted Infections (IUSTI) European Guidelines for syphilis management, lidocaine has been used as a diluent for BPG since 1998. In the United States (US), BPG often comes prepackaged and lidocaine is unable to be used as a diluent with the same ease as it is in Europe. In light of this, the investigators propose a randomized controlled trial of benzathine penicillin G with and without lidocaine to quantify any site pain reduction with lidocaine in patients being treated for syphilis.

This study is a randomized, double blinded, placebo controlled trial. During this study, patients needing BPG treatment for syphilis will be screened for any penicillin allergies and consented to their participation. Each participant will receive 2 injections of BPG, 1.2 million units each (2x1.2 million units = 2.4 million units, the standard dose for syphilis treatment), as intramuscular injections, one in each gluteal muscle, with one of the injections randomly having 0.5ml of 1% lidocaine added while the other has 0.5 ml normal saline solution. The side of each injection will be randomized by the medical assistant (MA)/nurse filling the vials and the injecting MA will be blinded, as well as the study participant, as to which vial contains lidocaine and which contains normal saline. The participants will then be asked to rate their pain from 0-10 on each site of injection at 10 minutes post injection, then again at 24 hours after injection via email electronic survey (via RedCap). The differences in pain from the two injections will be compared and analyzed to see if lidocaine reduces pain associated with BPG injections compared to the control of normal saline added to BPG.

DETAILED DESCRIPTION:
The purpose of the study is to test the question of: Does the addition of 0.5ml 1% lidocaine compared to 0.5 ml normal saline solution to 1.2 million units of benzathine penicillin G affect the pain experienced by individuals being treated for Treponema pallidum (syphilis) infections at 10 minutes and 24 hours post injection?

Background

Prior Literature and Studies, and Rationale for this Study

There is evidence to suggest that lidocaine can help reduce the pain associated with intramuscular injections of benzathine penicillin G or bicillin, used to treat syphilis infections. A study published in the Journal of Pediatric Infectious Diseases in 1998 found that the use of lidocaine as a diluent of BPG significantly reduced the pain of injection. Another study by Estrada et al in 2019 looked at the addition of 1% mepivicaine as diluent for PGB vs PGB alone and showed that mepivicaine significantly decreased pain experienced by participants. Per the IUSTI European Guidelines for Syphilis management, lidocaine is used as a diluent for benzathine penicillin G since 1998. No studies have been performed thus far looking at prefilled benzathine penicillin G syringes and the possibility of inserting lidocaine to the injection to decrease the pain experienced by individuals being treated for syphilis infections, instead of using lidocaine as a diluent which is not possible for the BPG formulations present here in the US.

Study Objectives

Primary Aim To see if there is any benefit of adding 0.5 ml 1% lidocaine to prepackaged Benzathine Penicillin G, with respect to pain, compared to standard of care, in the treatment of Treponema pallidum infections, both 10 minutes and 24 hours after injection.

Secondary Aim To see if there are any adverse effects of adding 0.5 ml 1% lidocaine to prepackaged Benzathine Penicillin G and to assess use of other pain medications 24 hours post injection.

Dose Rationale and Risk/Benefits Use of 0.5 ml 1% lidocaine was decided upon based off the size of the prefilled BPG syringe and the room for additional liquid within the syringe. 1% lidocaine is commonly used as a pain relief measure in clinical settings for injections and other procedures.

Overview or Design Summary This study is a double blinded randomized placebo control trial of addition of the effect on pain of the addition of 0.5ml 1% lidocaine solution to prepackaged benzathine Penicillin G injection, compared to addition of 0.5 ml normal saline solution, in adults being treated for syphilis (Treponema pallidum) infections, within the Infectious Diseases Clinic at Washington University in St. Louis.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or above
* Confirmed syphilis diagnosis (reactive RPR with confirmatory treponemal testing)
* Receiving first injection in series if patient requires 3x weekly injections for syphilis treatment

Exclusion Criteria:

* Penicillin allergy (anaphylaxis)
* Lidocaine allergy (anaphylaxis)
* Second or third injection in series if patient requires 3x weekly injections for syphilis treatment
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mean Pain Score (0-10) of Benzathine Penicillin G + Lidocaine Injection 10 minutes post injection | 10 minutes
  The average rating of participants' injection site pain with added lidocaine from 0 (no pain) to 10 (extreme pain) at 10 minutes post injection
Mean Pain Score (0-10) of Benzathine Penicillin G + Saline Injection 10 minutes post injection | 10 minutes
  The average rating of participants' injection site pain with added lidocaine from 0 (no pain) to 10 (extreme pain) at 10 minutes post injection
Relative difference of mean pain scores between injection types 10 minutes post injection | 10 minutes
  Comparative t-test of means of pain scores at injections sites at 10 minutes post injection
Mean Pain Score (0-10) of Benzathine Penicillin G + Lidocaine Injection 24 hours post injection | 24 hours
  The average rating of participants' injection site pain with added lidocaine from 0 (no pain) to 10 (extreme pain) at 24 hourspost injection
Mean Pain Score (0-10) of Benzathine Penicillin G + Saline Injection 24 hours post injection | 24 hours
  The average rating of participants' injection site pain with added lidocaine from 0 (no pain) to 10 (extreme pain) at 24 hours post injection
Relative difference of mean pain scores between injection types at 24 hours post injection | 24 hours
  Comparative t-test of means of pain scores at injections sites at 24 hours post injection

SECONDARY OUTCOMES:
Rate of Adverse reactions | 7 days
  To see if there are any adverse effects of adding 0.5 ml 1% lidocaine to prepackaged Benzathine Penicillin G
Rate of Use of other pain medications | 24 hours
  To assess use of other pain medications 24 hours post injection.

CONTACTS AND LOCATIONS:
Locations (1):
- WashU Infectious Diseases Clinic, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amir J, Ginat S, Cohen YH, Marcus TE, Keller N, Varsano I. Lidocaine as a diluent for administration of benzathine penicillin G. Pediatr Infect Dis J. 1998 Oct;17(10):890-3. doi: 10.1097/00006454-199810000-00008. PMID 9802630
- [Background] Janier M, Hegyi V, Dupin N, Unemo M, Tiplica GS, Potocnik M, French P, Patel R. 2014 European guideline on the management of syphilis. J Eur Acad Dermatol Venereol. 2014 Dec;28(12):1581-93. doi: 10.1111/jdv.12734. Epub 2014 Oct 27. PMID 25348878
- [Background] Estrada V, Santiago E, Cabezas I, Cotano JL, Carrio JC, Fuentes-Ferrer M, Vera M, Ayerdi O, Rodriguez C, Lopez L, Cabello N, Nunez MJ, Puerta T, Sagastagoitia I, Del Romero J. Tolerability of IM penicillin G benzathine diluted or not with local anesthetics, or different gauge needles for syphilis treatment: a randomized clinical trial. BMC Infect Dis. 2019 Oct 23;19(1):883. doi: 10.1186/s12879-019-4490-5. PMID 31646969

DOCUMENTS (2):
  • Study Protocol (2024-01-25): https://cdn.clinicaltrials.gov/large-docs/25/NCT06391125/Prot_000.pdf
  • Informed Consent Form (2024-01-25): https://cdn.clinicaltrials.gov/large-docs/25/NCT06391125/ICF_001.pdf